CLINICAL TRIAL: NCT06222307
Title: The Effects of Game-Based Exercises on Upper Extremity Muscle Strength, Sensory and Functionality: A Randomized Controlled Study
Brief Title: The Effects of Game-Based Exercises on Upper Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KARATAY_EAK
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-01

CONDITIONS: Development, Human
Keywords: Game-Based Exercises; Upper Extremity; Muscle Strength; Functionality

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: One (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Game-Based Exercises (Experimental): The participants will engage in game-based exercise training twice a week for a total of 6 weeks. Each session will last for 45 minutes, and to ensure participants' sustained engagement, the activities will vary weekly. Here's an outline of the weekly activities:
  Interventions: Other: Game-Based Exercises
- Control (No Intervention): No intervention will be applied to the control group

INTERVENTIONS:
Other: Game-Based Exercises — Week 1: Dough Kneading, Sorting Legumes, Cutting Lines with Scissors, Coloring with Dry Crayons Week 2: Dough Rolling, Scissor Use, Crumpling Paper, Finger Exercises, Tying Knots with Rubber Bands Week 3: Dough Cutting, Dough Rolling, Dough Stretching, Sewing with Needles, Wrapping Thread like a Spool, Sorting Legumes, Untying Knots in String Week 4: Rhythm Exercises, Dough Kneading and Rolling, Scissor Use, Sorting Legumes, Untying Knots in String Week 5: Stringing Beads on Thread, Unlocking, Tearing Paper, Sorting Legumes, Untying Knots in String Week 6: Tying Shoe Laces, Opening-Closing Jar Lids, Sorting Legumes
  Arms: Game-Based Exercises

SUMMARY:
The aim of this research is to investigate the impact of game-based exercises on upper extremity muscle strength, sensory perception, and functionality in adult individuals. The focus lies in measuring and assessing the effects of these exercises on this particular group. The goal is to determine the potential benefits of game-based exercises concerning upper extremity muscle strength, sensory perception, and overall functionality in adults.

DETAILED DESCRIPTION:
This study focuses on exploring how game-based exercises affect upper extremity muscle strength, sensory perception, and functionality in adults. It addresses the potential impact of these exercises on physical activity levels, sensory development, and body awareness. The research highlights the significance of physical engagement, particularly in digitally inactive environments, emphasizing the need for supportive physical activity interventions. Additionally, it delves into the intricate hand movements and functions related to grasping activities, emphasizing the importance of sensory perceptions in these processes. Ultimately, the study aims to understand the correlation between game-based exercises and various facets of upper extremity functionality in adults.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria comprise participants aged between 18 and 25 years, having good overall health with no significant upper extremity issues.
* Participants should demonstrate active use of both hands.
* Preference is given to individuals who have not previously engaged in regular upper extremity-focused exercises or do not have a habit of regular exercise.
* Voluntary participation in the study and willingness to comply with program requirements are necessary.

Exclusion Criteria:

* Encompass individuals with significant upper extremity disorders or a history of serious - hand, arm, or shoulder injuries,
* Those with sensory impairments,
* Individuals whose health conditions deem them unsuitable for participation in the exercise program,
* Individuals outside the specified age range,
* Participants who have previously engaged in upper extremity-focused exercise or similar studies

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Hand Muscle Strength Assessment | Baseline measurement before the Gamed-Based Exercises begin (pre-intervention), post-intervention at week 6
  Hand muscle strength will be evaluated with the Jamar Hand Dynamometer. The unit of measurement for evaluations is kilogram-force.
Finger Muscle Strength Assessment | Baseline measurement before the Gamed-Based Exercises begin (pre-intervention), post-intervention at week 6
  Pinch force will be measured with Jamar Hydraulic Pinchmeter. The unit of measurement for evaluations is kilogram-force.

SECONDARY OUTCOMES:
Sensory Assessment | Baseline measurement before the Gamed-Based Exercises begin (pre-intervention), post-intervention at week 6
  Sensory Assessment will be evaluated by two-point discrimination test. The unit of measurement for evaluations is milimeter.
Functional Assessment | Baseline measurement before the Gamed-Based Exercises begin (pre-intervention), post-intervention at week 6
  Functional assessment will be evaluated with the Nine Hole Peg Test. The unit of measurement for evaluations is seconds.

CONTACTS AND LOCATIONS:
Overall Officials: EMİNE ARSLAN KILIÇOĞLU, PhD(c), Principal Investigator — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No